CLINICAL TRIAL: NCT02677649
Title: Microbiota Diversity and Composition and Polyphenol Bioavailability: a Controlled Feeding Trial With a Plant Free Diet Containing Whole Cranberry Powder
Brief Title: Microbiota Diversity and Composition and Polyphenol Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Oliver Chen, Scientist I, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2870
Record Dates: First submitted 2016-02-03; First posted 2016-02-09 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Fecal Microbiota
Keywords: cranberry, microbiome, polyphenols, healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cranberry (Active Comparator): 30 grams/day freeze dried whole cranberry powder added to a basal diet comprising meats, dairy products, simple sugars, and stevia
  Interventions: Other: cranberry
- placebo (Placebo Comparator): 30 grams/day placebo powder [made with maltodextrin (CPC Maltrin M-180), citric acid, artificial cranberry flavor (Lorann oils), fructose, red color (Lorann oils), and grape shade] added to a basal diet comprising meats, dairy products, simple sugars, and stevia
  Interventions: Other: placebo

INTERVENTIONS:
Other: cranberry — the effect of cranberry on the gut microbiota
  Arms: cranberry
Other: placebo — the effect of placebo on the gut microbiota
  Arms: placebo

SUMMARY:
Composition and diversity of intestinal microbiota that are subject to the influence of diet have a significant impact on health in the gut and whole body via complex interactions between food constituents, bacteria, and host. Polyphenols are poorly absorbed in the upper gastrointestinal tract and reach the colon, where they may have a reciprocal relationship with microbiota. Because how polyphenols mediate gut health and reduce risk for other pathogenesis remains to be elucidated, we propose to conduct a pilot controlled feeding study to examine the impact of polyphenols and other constituents in the free dried whole cranberry powder (FWCP) on composition and diversity of gut microbiota, as well as to substantiate bioavailability of cranberry polyphenols. The central hypothesis underlying the proposed research is that FWCP polyphenols will diminish the magnitude of a plant food free diet induced increase in Alistipes, Bilophila and Bacteroides and will increase Enterococcus, Bifidobacterium, Eggerthella lenta, and Blautia coccoides-Eubacterium rectale groups. The proposed research is novel as no study has examined the specific impact of FWCP polyphenols incorporated into a plant food free diet on gut microbiota. This proposed study is innovative because the positive results will demonstrate with a high degree of confidence that the impact of FWCP constituents on production of beneficial short chain fatty acids, carcinogenic bile acids, and atherogenic trimethylamine. The results generated from the study using a plant food free dietary regimen as the background diet will provide definite proof on microbial modulating actions of FWCP, inform mechanism of actions in urinary tract infection (UTI), and be used to formulate messages in consumer communications for gut health.

DETAILED DESCRIPTION:
Investigators propose conducting a randomized, controlled feeding, crossover trial in 10 adults who have a regular bowel movement (≥5 times/wk) and are willing to consume a diet free of plant foods. The trial will include two 5-d intervention phases with a 2-wk washout period between crossovers. All meals will be provided to subjects during the intervention phases. Subjects will be randomly assigned to receive either Con or FWCP diet containing 30 gram matched placebo or FWCP. The dose is selected in order to provide sufficient amounts of flavonoid and PAC that can be comparable to the average flavonoid and PAC intake at 157 mg and 95 mg/d, respectively in US. The plant food free diet will be formulated to contain only animal based ingredients. All meals will be designed and overseen by Helen Rasmussen, PhD, RD, and be prepared in the kitchen of the Metabolic Research Unit. Packed frozen meals will be provided to subjects to consume at home or work. Coffee, tea, and other plant-based beverages will not be allowed during the intervention phases.

All subjects will be required to provide their informed consent prior to enrolling in the study. Individuals will be screened for study eligibility according to the exclusion criteria, as followed: 1) no antibiotic medications or drugs known to influence fecal microbiota were taken 3 mo before the study; 2) active treatment for doctor diagnosed diseases, such as cancer, cardiovascular diseases, gastrointestinal diseases; 3) regular use of any dietary supplements; 4) colonoscopy 2 mo prior to their enrollment or scheduled during the study; 5) values of standard blood biochemistries are critically abnormal based on study physician's discretion; and 6) use of ≥14/wk serving of alcohol. Subjects who meet all other eligibility criteria and have values of blood biochemistries within normal ranges will be asked to participate in the study.

During the trial, eligible subjects will be required to attend 1 screening visit and 9 study visits over 5-7 wks. At the end of Visits 2 and 6, subjects will receive the randomly assigned frozen meals and begin consuming the study meals for 5 d. Subjects may consume the study meals ≥5 da until the post-intervention stool sample is collected. The whole stool sample will be placed in a sealed bag and then in a cooler with ice packs and transported to the MRU within 24 h. Morning spot urine and 30 mL fasted blood as well as all other clinical data will be collected before and after each intervention phase. All collected samples will be stored at -80 degree C until uses.

The sample size of the human trial was estimated based on the effect of FWCP on the plant food free diet induced increase in bile tolerant bacteria and on the increase in Enterococcus, Bifidobacterium, Eggerthella lenta, and Blautia coccoides-Eubacterium rectale. Since there is no data in the literature illustrating the effect of FWCP on bile tolerant bacteria for power calculation, investigators will employ in the proposed crossover controlled feeding trial 10 subjects to test our hypothesis.

Fecal DNA will be extracted by enzymatic digestion and bead-beating steps followed by the use of QIAamp Stool DNA Mini Kit (Qiagen). 16S rRNA gene amplicons will be generated from the extracted DNA using PCR with a barcoded primer set targeted to the V4 variable region. Amplicons will be sequenced on an Illumina ® MiSeq Sequencer at the Tufts University Core Facility which is directed by Dr. Anne Kane. Microbiota Analysis will be performed using Qiime v 1.7. Operational taxonomic units will be generated using UClust. Alpha and beta diversity parameters will be calculated using Qiime. Urinary flavonoids and phenolic acids will be determined by our routine HPLC-electrochemical detection method. Anthocyanins and their glucuronidate metabolites in urine will be quantified by a LC-MS/MS assay investigators use routinely. Fecal short chain fatty acids will be determined using a GC-MS method that has been established in our laboratory. The pH value in the fecal water of the feces will be determined using a pH meter after centrifugation. Individual bile acids in feces will be determined using a LC-QTOF-MS method. TMA in feces will be determined using a spectrophotometric assay.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-55 y
2. BMI between 18.5-29.9 kg/m2
3. Bowel movement ≥3 times/wk
4. Consume ≥3 servings of fruits and vegetables daily on average
5. Willing to consume animal based diets for ≥10 days
6. Willing to consume freeze-dried whole cranberry powder
7. Willing to not take prebiotics and probiotics during the trial
8. Do not have allergic reaction to cranberries

Exclusion Criteria:

1. Colonoscopy 2 mo prior to their enrollment or scheduled during the study
2. No antibiotic medications or drugs known to influence fecal microbiota were taken or used 3 mo before the study
3. History of a bilateral mastectomy
4. History of autoimmune disorders (rheumatoid arthritis, lupus, multiple sclerosis, vitiligo, psoriasis)
5. Consume <3 servings of fruits and vegetables daily one average
6. Gastrointestinal diseases, conditions, or medications influencing gastrointestinal absorption including active peptic ulcer disease or inflammatory bowel disease which will be found based on the self-report during the screening visit
7. Regular use of any acid-lowering medications (≥3 times/week)
8. Use of ≥14/wk serving of alcohol (168 oz beer, 56 oz wine, 14 oz hard liquor)
9. Intend to be pregnant, pregnancy, and breastfeeding
10. Infrequent (<3/wk) or excessive (>3/d) number of regular bowel movements
11. Active treatment for cancer (except non-melanom skin cancer) and cardiovascular disease of any type >1 y
12. Having diabetes and/or receiving medications for diabetic condition, which will be found based on the self-report during the screening visit
13. Thyroid disease unstable or medication adjustments in past 6 months, which will be found based on the self-report during the screening visit
14. Values of standard blood biochemistries are unacceptable for the study based on study physician's discretion
15. vegetarians and vegans, unwillingness or inability to consume animal-based foods including chicken, turkey, beef, eggs, cheese, other milk products, etc. Allergy to eggs or milk/dairy products.
16. Use anticoagulants, such as heparin, warfarin (coumadin) in past 6 months
17. On or planning to be on a weight loss regimen
18. Regular use of any dietary supplements containing vitamins, minerals, herbal or other plant-based preparations, fish oil supplements (including cod liver oil) or homeopathic remedies; however, subjects who are willing to refrain from the use of these supplements at enrollment and throughout the entire study may be considered eligible
19. Use of monoamine oxidase inhibitors (MAOIs)
20. Glomerular filtration rate (GFR) <60 mL/min/1.73 m2
21. Total cholesterol (TC) >250 mg/dL
22. Total triglycerides (TG) >300 mg/dL

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
fecal microbiome | The change in fecal microbiome after consuming the intervention diets for 5 days.
  16S rRNA in feces will be determined to profile microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Chen, PhD, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging, Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No